CLINICAL TRIAL: NCT00205231
Title: A Pilot Study to Examine the Feasibility and Effect on Tumor Necrosis Factor (TNF) Inhibition on HIV Disease
Brief Title: A Pilot Study to Examine the Feasibility and Effect of Tumor Necrosis Factor (TNF) Inhibition on HIV Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Immunex Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2001-557
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: HIV Infections
Keywords: HIV
MeSH Terms: conditions — HIV Infections | interventions — Etanercept

INTERVENTIONS:
Drug: etanercept

SUMMARY:
This pilot study will investigate the safety and effect of etanercept in HIV infection by studying HIV replication and immune function (as measured by CD4 counts) in individuals with HIV infection.

ELIGIBILITY:
Inclusion Criteria:

* Adults greater than 18 years of age with documented HIV infection
* Highly active antiretroviral therapy (HAART) regimens as defined by the Department of Health and Human Services guidelines; stable regimens for 12 weeks.
* CD4 greater than 200 at time of study enrollment
* Stable monitoring labs (hematology survey with differential, ALT, creatinine)
* Absolute neutrophil count within normal limits

Exclusion Criteria:

* AIDS defining illness within the last 6 months
* Acute bacterial, viral, or fungal infection within the last 1 month, or history of recurring infections
* Women who are pregnant or nursing
* Hypersensitivity to etanercept
* Previous use of etanercept
* Acute malignancy in the last 5 years excluding in situ cervical cancer (CA) and common skin cancers (non melanoma)
* History of active or latent tuberculosis
* History of demyelinating nerve disease
* History of seizure disorder
* Latex allergy
* Subject has any of the following laboratory values within 30 days of baseline:

  * hemoglobin concentration < 10.0 g/dl for men and < 9.0 g/dl for women
  * platelet count < 75,000/mm3
  * AST or ALT > 5x upper limit of normal (ULN)
  * serum creatinine > 2.5x ULN
  * serum pancreatic amylase > 1.5 ULN
* Subject requiring treatment with immunomodulating agents, such as systemic corticosteroids, interleukins, vaccines, or interferon
* Subjects who chronically use any over-the-counter (OTC) or prescription medication (except vitamins) must not change the regimen or switch their medication within 3 days of drug administration and until discharged from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2002-05; Primary Completion 2004-05-01 (Actual); Study Completion 2004-05-01 (Actual)

PRIMARY OUTCOMES:
changes in CD4 counts
changes in HIV-RNA levels

SECONDARY OUTCOMES:
development of infections
degree of TNF inhibition by measuring TNF levels
changes in hematologic and biochemical laboratory tests

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Urban, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States